CLINICAL TRIAL: NCT05358678
Title: Cesarean Section Scar Niche: The Impact on Assisted Reproductive Technology Outcome
Brief Title: Cesarean Section Scar Niche: The Impact on ART Outcome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rahem Fertility Center (Other)
Collaborators: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Eman Elgindy, Professor of obstetrics and Gynecology Zagazig University Faculty of Medicine, Rahem Fertility Center
Other Study IDs: 9385
Record Dates: First submitted 2022-03-22; First posted 2022-05-03 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Cesarean Section; ART
Keywords: Cesarean Section niche; ART

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases with cs niche: 133 cases with cs niche undergoing ART will be included. Pituitary suppression will be achieved by long or antagonist protocol. For long protocol, GnRH agonist will be administered for 10-14 days starting from mid-luteal phase of preceding cycle. After confirmation of down regulation, gonadotropins will be given from second or third day of cycle in a daily dose of (150-300 IU). Gonadotropins therapy will be tailored according to age, BMI, antral follicle count, antimullerian hormone and previous response. In antagonist protocol, gonadotropins will be given from second or third day of cycle in a daily dose of (150-300 IU). GnRH antagonist will be adjusted according to patient response. On the 5th -6th day of stimulation, sonography will be performed and repeated every 1-3 days with regular estradiol assessment. When at least 3 follicles reach ≥ 17 mm in mean diameter, trigger will be given. Oocytes pick up will be performed 34-36 hour after triggering.
  Interventions: Diagnostic Test: cs niche group
- cases without cs niche: 133 cases without cs niche undergoing ART will be included. Pituitary suppression will be achieved by long or antagonist protocol. For long protocol, GnRH agonist will be administered for 10-14 days starting from mid-luteal phase of preceding cycle. After confirmation of down regulation, gonadotropins will be given from second or third day of cycle in a daily dose of (150-300 IU). Gonadotropins therapy will be tailored according to age, BMI, antral follicle count, antimullerian hormone and previous response. In antagonist protocol, gonadotropins will be given from second or third day of cycle in a daily dose of (150-300 IU). GnRH antagonist will be adjusted according to patient response. On the 5th -6th day of stimulation, sonography will be performed and repeated every 1-3 days with regular estradiol assessment. When at least 3 follicles reach ≥ 17 mm in mean diameter, trigger will be given. Oocytes pick up will be performed 34-36 hour after triggering.

INTERVENTIONS:
Diagnostic Test: cs niche group — A niche is formally defined by the European Niche Taskforce as an indentation of the uterine myometrium of at least 2 mm at the site of the CS scars. A niche can be sub classified as follows:
  1. Simple niche
  2. Simple niche with one branch
  3. Complex niche (with more than one branch).
  The following measurements will be taken:
  * Length.
  * Depth.
  * Width.
  * RMT (residual myometrium thickness).
  * AMT (adjacent myometrium thickness).
  * Distance between the niche and the VV (vesico-vaginal) fold.
  * Distance between the niche and the external os. We will also comment on the position of the uterus (AVF or RVF), presence or absence of intra cavitary fluid and its thickness.
  Groups: cases with cs niche

SUMMARY:
To evaluate the impact of the presence of cesarean section niche and its characteristics on the outcome of ART cycles.

DETAILED DESCRIPTION:
The incidence of Cesarean section (CS) is increasing worldwide, with a corresponding increase in its associated complications. The well-known complications are infection, hemorrhage, and increased risk of obstetric complications in subsequent pregnancies, like morbidly adherent placenta, cs scar pregnancies and uterine rupture.

In addition, some studies emphasize the effect of cesarean sections on reduced fertility. A meta-analysis reported that a Caesarean section reduces the probability of subsequent pregnancy by 10%, compared with a previous vaginal delivery.

The cesarean section niche is defined as an indentation of the uterine myometrium of at least 2 mm at the site of the caesarean scar. The most common symptom of niche is abnormal uterine bleeding. Meanwhile, other symptoms include dysmenorrhea, chronic pelvic pain, dyspareunia, and sub-fertility/infertility.

The detection of a cesarean section niche depends on the operator and the diagnostic method used. This can be 2D, 3D transvaginal sonography, sonohysterography or hysteroscopy.

Regarding ART, the presence of cs niche was reported to reduce the chances of embryo implantation, and increase the rate of spontaneous miscarriages, especially if the implantation is close to it or in the niche.

The presence of a niche may increase the difficulty of embryo transfer procedure, clinicians need to be aware of its presence and the transfer should be done under ultrasound guidance to ensure the catheter bypasses the niche and enters the uterine cavity.

Still the impact of c.s niche and its characteristics on outcome of ART is not clear.

ELIGIBILITY:
Inclusion criteria:

1. Aged from 18 - 37 years old.
2. Having a history of one or more previous CS with ultrasonographic visible cesarean section niche (for the group with cs scar niche), which is regarding to European Niche Taskforce is an indentation of the uterine myometrium of at least 2 mm at the site of the CS scar (Jordans et al., 2019).
3. A normal uterus with no anomalies or pathologies.
4. At least one good-quality embryo available for transfer.

Exclusion criteria:

1. Younger than 18 or older than 37 years old.
2. Congenital uterine abnormality or pathology.
3. Presence of a hydrosalpinx.
4. ICSI cycles with TESE samples.

Ages: 18 Years to 37 Years | Sex: Female
Age Groups: Adult
Study Population: It will be carried out in the department of Obstetrics and Gynecology, Zagazig University and in Rahem fertility center
Sampling Method: Non-Probability Sample
Enrollment: 266 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
The effect of cesarean scar niche and its characteristics on ongoing pregnancy rate of ART cycles. | 3 months
  Ongoing pregnancy: defined as a viable intrauterine pregnancy of at least 12 weeks duration confirmed on an ultrasound scan

SECONDARY OUTCOMES:
Clinical pregnancy | 6 weeks
  Clinical pregnancy: A pregnancy diagnosed by ultrasonographic visualization of one or more gestational sacs.

CONTACTS AND LOCATIONS:
Overall Officials: Eman Elgindy, MD, PhD, Principal Investigator — Rahem Fertility Center
Locations (1):
- Rahem Fertility Center, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schepker N, Garcia-Rocha GJ, von Versen-Hoynck F, Hillemanns P, Schippert C. Clinical diagnosis and therapy of uterine scar defects after caesarean section in non-pregnant women. Arch Gynecol Obstet. 2015 Jun;291(6):1417-23. doi: 10.1007/s00404-014-3582-0. Epub 2014 Dec 17. PMID 25516174
- [Background] Clark EA, Silver RM. Long-term maternal morbidity associated with repeat cesarean delivery. Am J Obstet Gynecol. 2011 Dec;205(6 Suppl):S2-10. doi: 10.1016/j.ajog.2011.09.028. Epub 2011 Oct 6. PMID 22114995
- [Background] D'Antonio F, Timor-Tritsch IE, Palacios-Jaraquemada J, Monteagudo A, Buca D, Forlani F, Minneci G, Foti F, Manzoli L, Liberati M, Acharya G, Cali G. First-trimester detection of abnormally invasive placenta in high-risk women: systematic review and meta-analysis. Ultrasound Obstet Gynecol. 2018 Feb;51(2):176-183. doi: 10.1002/uog.18840. PMID 28833750
- [Background] Gurol-Urganci I, Bou-Antoun S, Lim CP, Cromwell DA, Mahmood TA, Templeton A, van der Meulen JH. Impact of Caesarean section on subsequent fertility: a systematic review and meta-analysis. Hum Reprod. 2013 Jul;28(7):1943-52. doi: 10.1093/humrep/det130. Epub 2013 May 3. PMID 23644593
- [Background] Jordans IPM, de Leeuw RA, Stegwee SI, Amso NN, Barri-Soldevila PN, van den Bosch T, Bourne T, Brolmann HAM, Donnez O, Dueholm M, Hehenkamp WJK, Jastrow N, Jurkovic D, Mashiach R, Naji O, Streuli I, Timmerman D, van der Voet LF, Huirne JAF. Sonographic examination of uterine niche in non-pregnant women: a modified Delphi procedure. Ultrasound Obstet Gynecol. 2019 Jan;53(1):107-115. doi: 10.1002/uog.19049. PMID 29536581
- [Background] Sandall J, Tribe RM, Avery L, Mola G, Visser GH, Homer CS, Gibbons D, Kelly NM, Kennedy HP, Kidanto H, Taylor P, Temmerman M. Short-term and long-term effects of caesarean section on the health of women and children. Lancet. 2018 Oct 13;392(10155):1349-1357. doi: 10.1016/S0140-6736(18)31930-5. PMID 30322585
- [Background] Ludwin A, Martins WP, Ludwin I. Evaluation of uterine niche by three-dimensional sonohysterography and volumetric quantification: techniques and scoring classification system. Ultrasound Obstet Gynecol. 2019 Jan;53(1):139-143. doi: 10.1002/uog.19181. No abstract available. PMID 30039641
- [Background] Naji O, Wynants L, Smith A, Abdallah Y, Saso S, Stalder C, Van Huffel S, Ghaem-Maghami S, Van Calster B, Timmerman D, Bourne T. Does the presence of a Caesarean section scar affect implantation site and early pregnancy outcome in women attending an early pregnancy assessment unit? Hum Reprod. 2013 Jun;28(6):1489-96. doi: 10.1093/humrep/det110. Epub 2013 Apr 12. PMID 23585560
- [Background] Lawrenz B, Melado L, Garrido N, Coughlan C, Markova D, Fatemi H. Isthmocele and ovarian stimulation for IVF: considerations for a reproductive medicine specialist. Hum Reprod. 2020 Jan 1;35(1):89-99. doi: 10.1093/humrep/dez241. PMID 31885047